CLINICAL TRIAL: NCT01028014
Title: Medication Effects on Periurethral Sensation, Urethral Sphincter Activity and Pressure Flow Parameters
Brief Title: Medication Effects on Periurethral Sensation,Urethral Sphincter Activity and Pressure Flow Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Holly Richter, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: VESI-9E03-UAB
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Results first posted 2011-09-05 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Urethral Sphincter Activity
MeSH Terms: interventions — Pseudoephedrine; Tamsulosin; Imipramine; cyclobenzaprine; Lactose; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Pseudoephedrine (Active Comparator): Pseudoephedrine 120mg extended release tablets
  Interventions: Drug: Pseudoephedrine
- Solifenacin (Active Comparator): Solifenacin 5mg capsule
  Interventions: Drug: Solifenacin
- Tamsulosin (Active Comparator): Tamsulosin 0.4mg capsule
  Interventions: Drug: Tamsulosin
- Imipramine (Active Comparator): Imipramine 25mg tablet
  Interventions: Drug: Imipramine
- Cyclobenzaprine (Active Comparator): Cyclobenzaprine 10mg tablet
  Interventions: Drug: Cyclobenzaprine
- Lactose capsules (Placebo Comparator): Sham
  Interventions: Drug: Lactose capsule

INTERVENTIONS:
Drug: Pseudoephedrine — Pseudoephedrine ER 120 mg by mouth once daily for 2 weeks
  Arms: Pseudoephedrine
Drug: Tamsulosin — Tamsulosin 0.4mg by mouth daily for 2 weeks
  Other Names: Flomax
  Arms: Tamsulosin
Drug: Imipramine — Imipramine 25mg daily by mouth for 2 weeks
  Other Names: Tofranil
  Arms: Imipramine
Drug: Cyclobenzaprine — Cyclobenzaprine 10mg daily by mouth for 2 weeks
  Other Names: Flexeril
  Arms: Cyclobenzaprine
Drug: Lactose capsule — Lactose capsule 1 by mouth daily for 2 weeks
  Arms: Lactose capsules
Drug: Solifenacin — Solifenacin 5mg by mouth daily for 2 weeks
  Other Names: VESIcare
  Arms: Solifenacin

SUMMARY:
Lower urinary tract symptoms such as urinary leakage and overactive bladder affect millions of American women. Women may develop these problems because the innervation of the muscles of the bladder and urethra are injured. Most research on treating these problems has focused on the abnormalities of the bladder muscle, but newer studies have shown abnormalities in the innervation and muscle function of the urethra.

Women with these symptoms may benefit from treatment with medications to improve their urethral function. However, to truly understand what types of medications will help women with these symptoms, the investigators wish to study how these medications affect innervation and muscle function in healthy women who do not have lower urinary tract symptoms.

DETAILED DESCRIPTION:
Women without urinary incontinence or bladder symptoms (healthy controls)will undergo urethral testing prior to randomization to one of 5 medications or placebo. Participants will take an oral medication for 2 weeks and then return for repeat testing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Females only
* Ages 19-51 and up including pre-menopausal older women who have had a normal menstrual cycle for the prior 3 months
* Able to take oral medication for 2 weeks
* For women of child bearing potential,willing to use an approved method of birth control during the study

Exclusion Criteria:

* Urinary Incontinence or other bladder symptoms
* Known neurologic disease that may impair urethral tone or sensation
* Currently taking a class of medication that is being tested (alpha-antagonists, anticholinergics, sympathomimetics, tricyclic antidepressants, or skeletal muscle relaxants)
* History of QTc prolongation or cardiac arrhythmia
* Pregnant, breastfeeding, or are less than 6 months postpartum
* Known hypersensitivity to or other contraindications to taking any of the study medications

Ages: 19 Years to 51 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly E Richter, PhD, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, The Kirklin Clinic, Birmingham, Alabama, United States

REFERENCES:
- [Result] Greer WJ; Gleason J; Szychowski JM; Goode P; Kenton K; Richter HE. Medication Effects on Urethral Current Perception Thresholds and Pressure Flow Parameters. Fem Pelv Med Recons Surg 2011;17:S33.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy women,ages 19-51 and up including pre-menopausal older women who have had a normal menstrual cycle for the prior 3 months.Participants were recruited via local newspaper. The first participant was enrolled 5/27/10. Recruitment ended August 31, 2010
Groups:
- Pseudoephedrine 120mg ER Daily: 120 mg extended release tablet one daily for 14 days
- Solifenacin 5mg Daily: 5 mg capsule, one daily for 14 days
- Tamsulosin 0.4mg Daily: 0.4 mg capsule, one daily for 14 days
- Imipramine 25mg Daily: 25 mg tablet, one daily for 14 days
- Cyclobenzaprine 10mg Daily: 10 mg tablet, one daily for 14 days
- Lactose Capsules, One Daily: sham lactose capsules, one daily for 14 days
Period: Overall Study
Arm/Group | Pseudoephedrine 120mg ER Daily | Solifenacin 5mg Daily | Tamsulosin 0.4mg Daily | Imipramine 25mg Daily | Cyclobenzaprine 10mg Daily | Lactose Capsules, One Daily
Started | 10 | 10 | 10 | 10 | 10 | 6
Completed | 9 | 8 | 10 | 9 | 9 | 4
Not Completed | 1 | 2 | 0 | 1 | 1 | 2
Not completed — Lost to Follow-up | 1 | 2 | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Pseudoephedrine 120mg ER Daily: 120 mg extended release, 1 daily for 14 days
- Solifenacin 5mg Daily: 5 mg capsule, 1 daily for 14 days
- Tamsulosin 0.4mg Daily: 0.4 mg capsule, 1 daily for 14 days
- Imipramine 25mg Daily: 25 mg tablet, 1 daily for 14 days
- Cyclobenzaprine 10mg Daily: 10 mg tablet, 1 daily for 14 days
- Lactose Capsules, One Daily: sham lactose capsules, 1 daily for 14 days
- Total: Total of all reporting groups
Arm/Group | Pseudoephedrine 120mg ER Daily | Solifenacin 5mg Daily | Tamsulosin 0.4mg Daily | Imipramine 25mg Daily | Cyclobenzaprine 10mg Daily | Lactose Capsules, One Daily | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 6 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 10 | 10 | 6 | 56
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Full Range); unit: years] | 36.6 [24 to 49] | 31.6 [21 to 35] | 35.5 [21 to 49] | 33.1 [21 to 50] | 38 [24 to 53] | 28.7 [21 to 35] | 34.3 [19 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 10 | 10 | 10 | 6 | 56
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 10 | 10 | 6 | 56

OUTCOME MEASURES:

1. Primary Outcome: Difference (Pre - Post) in Amplitude (Microvolts) of Urethral Sphincter Activity as Measured by Quantitative Concentric Needle EMG
Description: Concentric needle EMG was used to measure urethral sphincter activity at 2-3 sites around the urethral meatus before and after 2 weeks of therapy with one of 6 randomly assigned medications. Two methods of quantitative electromyography were performed on all subjects. (1) Multi-Motor Unit Action Potential (MUP) analysis, which has been shown to be the most sensitive technique in distinguishing neuropathic from control muscles; and (2) interference pattern analysis (IPA) which reflects changes in MUP recruitment from weak effort to maximal contraction.
Time Frame: 2 weeks
Population: The planned number of participants was per protocol based on power calculation. Actual number may differ based on withdrawal from the study or loss to follow-up.Participants randomized to Pseudoephedrine 120 mg ER,Solifenacin 5 mg, Tamsulosin 0.4mg, Imipramine 25mg, Cyclobenzaprine 10 mg, or a sham Lactose capsule, 1 a day for 14 days.
Measure: Median (Inter-Quartile Range); unit: microvolts
Groups:
- Pseudoephedrine 120mg ER Daily: 120 mg extended release, 1 tablet daily for 14 days
- Solifenacin 5mg Daily: 5 mg capsule, 1 capsule daily for 14 days
Arm/Group | Pseudoephedrine 120mg ER Daily | Solifenacin 5mg Daily | Tamsulosin 0.4mg Daily | Imipramine 25mg Daily | Cyclobenzaprine 10mg Daily | Lactose Capsules, One Daily
Number analyzed (Participants) | 8 | 8 | 10 | 9 | 9 | 4
microvolts | -18 [-108 to 89] | 10 [-56 to 60] | 11 [-102 to 52] | -15 [-157 to 75] | 12 [-71 to 104] | 36 [23 to 45]
Statistical Analysis 1: Comparison: Pseudoephedrine 120mg ER Daily vs Solifenacin 5mg Daily vs Tamsulosin 0.4mg Daily vs Imipramine 25mg Daily vs Cyclobenzaprine 10mg Daily vs Lactose Capsules, One Daily; Using difference in EMG amplitude as primary outcome, assuming standard deviation of 6, we had greater than 80% power to detect a 10-microvolt change in urethral muscle activity with sample size of 9 participants per group. Due to non-normality and small sample sizes, non-parametric tests were used and data presented as median (IQR). Kruskal-Wallis p-values are reported to compare median scores across groups. Wilcoxon sign-test p-values are reported to evaluate 2-week change within groups; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — P values comparing differences across groups, as well as within group changes, were all >0.05.P-values were not adjusted for multiple testing; p<0.05 was considered statistically significant

2. Other Pre Specified Outcome: Difference (Pre - Post) in Urethral Sensation (Milliamps) as Measured by Current Perception Threshold Testing.
Description: Current Perception Threshold testing was used to measure urethral sensation before and after 2 weeks of therapy with one of 6 randomly assigned medications. We performed CPT testing in the urethra using a Neurometer®, which is a constant current stimulator capable of delivering sine wave electrical stimuli at 3 frequencies (2000 Hz, 250 Hz and 5 Hz). At all 3 frequencies, the stimulus intensity was gradually increased until first perceived, and then decreased until no longer perceptible. CPT values were obtained using a semi-automated forced choice paradigm.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Milliamps
Arm/Group | Pseudoephedrine 120mg ER Daily | Solifenacin 5mg Daily | Tamsulosin 0.4mg Daily | Imipramine 25mg Daily | Cyclobenzaprine 10mg Daily | Lactose Capsules, One Daily
Number analyzed (Participants) | 8 | 8 | 10 | 9 | 9 | 4
Milliamps | 0.06 [0.0 to 0.68] | 0.06 [-0.01 to 0.34] | -0.8 [-0.8 to 0.04] | -0.12 [-0.4 to 0.12] | 0.0 [-0.16 to 0.28] | 0.03 [-0.03 to 0.05]
Statistical Analysis 1: Comparison: Pseudoephedrine 120mg ER Daily vs Solifenacin 5mg Daily vs Tamsulosin 0.4mg Daily vs Imipramine 25mg Daily vs Cyclobenzaprine 10mg Daily vs Lactose Capsules, One Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

3. Other Pre Specified Outcome: Difference (Pre - Post) in Maximum Urine Flow Rate (Qmax) (Milliliters Per Second) as Measured by Pressure Flowmetry
Description: Pressure Flowmetry was used to measure maximum urine flow rate (Qmax)before and after 2 weeks of therapy with one of 6 randomly assigned medications. A 300 cc bladder fill was performed through the catheter, the catheter was removed, and transurethral and transrectal pressure transducers were placed for the pressure flow study. Voiding was performed in the seated position. Information obtained for the database included Qmax, average flow rate, time to Qmax, detrusor pressure at maximum flow rate, voided volume, and a calculated post-void residual.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: milliliters per second
Arm/Group | Pseudoephedrine 120mg ER Daily | Solifenacin 5mg Daily | Tamsulosin 0.4mg Daily | Imipramine 25mg Daily | Cyclobenzaprine 10mg Daily | Lactose Capsules, One Daily
Number analyzed (Participants) | 8 | 8 | 10 | 9 | 9 | 4
milliliters per second | -7.3 [-23.8 to 7.2] | 5.0 [-24.5 to 21.4] | -5.6 [-45.3 to 16.5] | -6.6 [-55.1 to 8.7] | 10.3 [-30.1 to 31.9] | 10.4 [-27.6 to 22.8]

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected from 5/27/10, the date of first participant enrolled, until 9/20/10 when the last participant completed the study.
Groups:
- Pseudoephedrine 120mg ER Daily: 120mg extended release, one daily for 14 days
- Cyclobenzaprine 10mg Daily: 10mg tablet, one daily for 14 days
Arm/Group | Pseudoephedrine 120mg ER Daily | Solifenacin 5mg Daily | Tamsulosin 0.4mg Daily | Imipramine 25mg Daily | Cyclobenzaprine 10mg Daily | Lactose Capsules, One Daily
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/6
Other Adverse Events (participants affected / at risk) | 2/10 | 1/10 | 1/10 | 2/10 | 0/10 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pseudoephedrine 120mg ER Daily (N=10) | Solifenacin 5mg Daily (N=10) | Tamsulosin 0.4mg Daily (N=10) | Imipramine 25mg Daily (N=10) | Cyclobenzaprine 10mg Daily (N=10) | Lactose Capsules, One Daily (N=6)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Dry mouth resolved after the first two days of study medication.
Headaches (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Reported migraine like headaches over the weekend. Headaches stopped two days later. No further problems with headaches.
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Subject had mild nausea at bedtime after taking study medication. Instructed to take medication iwth food at dinner time and the problem was resolved.
Vaginal Yeast Infection (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Problem resolved after she took Diflucan that she had at home.
Voiding discomfort (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Discomfort with voiding; improved with Azo-Standard.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No